CLINICAL TRIAL: NCT03102515
Title: Transversus Abdominis Plane Block vs Continuous Infiltration Wound Catheter for Analgesia After Caesarean Section: a Randomized Trial. (TAP-CAT Study)
Brief Title: Transversus Abdominis Plane Block vs Continuous Infiltration Wound Catheter for Analgesia After Caesarean Section
Acronym: TAP-CAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Purpose: Treatment
Other Study IDs: 2016-A00131-50
Record Dates: First submitted 2017-03-31; First posted 2017-04-05 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal-anesthesia (Other): Caesarean section performed under spinal anaesthesia and receiving either USG-TAP block or CIC
  Interventions: Drug: USG-TAP block; Drug: CIC
- Epidural-anesthesia (Other): Caesarean section performed under epidural anaesthesia and receiving either USG-TAP block or CIC
  Interventions: Drug: USG-TAP block; Drug: CIC

INTERVENTIONS:
Drug: USG-TAP block
Drug: CIC

SUMMARY:
Analgesia following surgery associates different intra-venous or oral analgesic drugs and sometimes opioids. To reduce opioid consumption, loco-regional anaesthesia might be administered as a complement. In the specific context of caesarean sections, pain control is mandatory to enable the mother to take care of her offspring and shorten their hospital stay. This intervention is mainly performed under neuraxial anaesthesia (spinal or epidural), enabling the injection of morphine in the subdural or epidural space, as part of a multimodal analgesia regimen.

Studies have evaluated continuous wound infiltration catheters (CIC) and ultrasound-guided (UGD) transabdominis plane (TAP) block, and both techniques and both techniques reduce postoperative morphine consumption. Recent studies have compared the two techniques and found conflicting results. Furthermore, they did not consider caesarean section performed under epidural analgesia, with a different neuraxial injection site, neither did they compared pain after postoperative day 2.

Consequently, the aim of this study was to compare resting and standing pain up to postoperative day 3 after caesarean section performed under spinal or epidural anaesthesia and receiving either USG-TAP block or CIC. Baseline hypothesis was that the continuous infiltration provided a better analgesia at day 2.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent,
* Age>/=18 years,
* Caesarean section under spinal or epidural anaesthesia
* Technique surgical "Cohen Stark méthod".

Exclusion Criteria:

* Patient refusal,
* Patient under guardianship,
* Contraindication to one of the two techniques,
* Cesarean section under general anesthesia
* Allergies to local anesthetics
* Maternal instability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-05-29 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-10-26 (Actual)

PRIMARY OUTCOMES:
Postoperative standing pain at day 2 | Evaluate standing pain at 48 hours postoperatively
  Assessment of Pain on Mobilization by a Numeric Scale of Pain

SECONDARY OUTCOMES:
standing and resting pain measured during the first 3 days | Evaluate pain at during 3 days postoperatively
  Assessment of Pain by a Numeric Scale of Pain
Cumulative dose of Tramadol during the first 3 days | during the first 3 days
Cumulative dose of nefopam during the first 3 days | during the first 3 days
Cumulative dose of oxycodone during the first 3 days | during the first 3 days
patient comfort assessed daily by visual analogic scale | during the first 3 days
  by visual analogic scale